CLINICAL TRIAL: NCT01670383
Title: Repository for Samples Collected From Sepsis and Postresuscitation Patients in Emergency Intensive Care Unit
Brief Title: Repository for Sepsis and Postresuscitation Samples
Status: Recruiting | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Gil Joon Suh, Professor, Seoul National University Hospital
Other Study IDs: SNUHEM-Repository-12-0001
Record Dates: First submitted 2012-08-08; First posted 2012-08-22 (Estimated); Last update posted 2023-11-24 (Actual); Status verified 2023-11

CONDITIONS: Cardiac Arrest; Sepsis
Keywords: Cardiac Arrest; Sepsis; Biological Markers; Anti-Inflammation Agents; Antioxidants
MeSH Terms: conditions — Heart Arrest; Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Patients sera at ICU admission, day-1, day-3 and day-7 are stored in deep freezer.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Postresuscitation group: Adults (age over 16 years old) who have survived from nontraumatic cardiac arrest and admitted to ICU.
- Sepsis group: Adults (age over 16 years old) who satisfy the sepsis criteria (SIRS>=2 and infection is suspected for a cause) and admitted to the ICU.

SUMMARY:
The objective of this study is to find a new therapeutic strategy by investigating the serial serum samples of patients with sepsis or postresuscitation state.

ELIGIBILITY:
Inclusion Criteria:

* Age over 16 years old
* Admitted to ICU
* Diagnosed as having sepsis or as postresuscitation status
* Definition of sepsis: 2 or more SIRS criteria + infection is suspected
* Definition of postresuscitation status: Survived from non-traumatic cardiac arrest

Exclusion Criteria:

* refusal to participate
* DNAR status

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Sepsis patients admitted to ICU Postresuscitation patients admitted to ICU
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2006-07; Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
1-month mortality | 1 month
  All cause mortality within 1-month

SECONDARY OUTCOMES:
Hospital mortality | until hospital discharge, an expected average of 2 weeks
  All cause mortality during hospitalization
ICU length of stay | Until ward transfer or discharge, an expected average of 7 days
Favorable neurologic outcome | at discharge, an expected average of 2 weeks and at 6-month
  Favorable neurologic outcome is used for outcome measure in postresuscitation patients only.
  Favorable neurologic outcome means cerebral performance category 1 and 2. This outcome is measured at discharge and 6-month after admission.

CONTACTS AND LOCATIONS:
Overall Officials: Gil Joon Suh, Professor, Study Director — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

REFERENCES:
- [Background] Angus DC, Linde-Zwirble WT, Lidicker J, Clermont G, Carcillo J, Pinsky MR. Epidemiology of severe sepsis in the United States: analysis of incidence, outcome, and associated costs of care. Crit Care Med. 2001 Jul;29(7):1303-10. doi: 10.1097/00003246-200107000-00002. PMID 11445675
- [Background] Dombrovskiy VY, Martin AA, Sunderram J, Paz HL. Rapid increase in hospitalization and mortality rates for severe sepsis in the United States: a trend analysis from 1993 to 2003. Crit Care Med. 2007 May;35(5):1244-50. doi: 10.1097/01.CCM.0000261890.41311.E9. PMID 17414736
- [Background] Cohen J. The immunopathogenesis of sepsis. Nature. 2002 Dec 19-26;420(6917):885-91. doi: 10.1038/nature01326. PMID 12490963
- [Background] Schneider A, Bottiger BW, Popp E. Cerebral resuscitation after cardiocirculatory arrest. Anesth Analg. 2009 Mar;108(3):971-9. doi: 10.1213/ane.0b013e318193ca99. PMID 19224811
- [Derived] Kim KS, Suh GJ, Jin M, Kwon WY, Jung YS, Kim T, Kim YT, Kim H, Park H. SECRETED TRYPTOPHANYL-tRNA SYNTHETASE 1 IS A PROGNOSTIC MARKER IN SEPSIS PATIENTS WITHOUT MONOCYTOPENIA. Shock. 2024 Jan 1;61(1):55-60. doi: 10.1097/SHK.0000000000002259. Epub 2023 Oct 20. PMID 37878497